CLINICAL TRIAL: NCT03967587
Title: Evaluation of Intravascular Monitoring of Partial PRessure of Oxygen for Neonatal intensiVE Care Patients
Acronym: IMPROVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The clinical investigation IMPROVE has been closed after a decision by the Swedish Medical Products Agency that the trial must comply to the new European medical regulation MDR.
Sponsor: Neosense Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IMPROVE
Record Dates: First submitted 2019-05-10; First posted 2019-05-30 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Catheters; Oxygen Saturation; Newborn, Infant, Disease
Keywords: Neonatal; Umbilical Arteries; Umbilical Veins; Oxygen Partial Pressure
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neosense Umbilical Catheter (Experimental)
  Interventions: Device: Neosense Umbilical Catheter

INTERVENTIONS:
Device: Neosense Umbilical Catheter — The Neosense umbilical catheter is used instead of the routinely used umbilical catheter

SUMMARY:
The study is a non-blinded trial with one single intervention in sick newborn infants. The Neosense umbilical catheter will be used instead of the routinely used umbilical catheter on infants where the treating physician has ordered use of an umbilical catheter. The catheter will be connected to the Neosense monitor/measuring unit.

Blood samples for blood gas analysis are collected from the patients according to the clinical routine (every 4th to 6th hour). Oxygen tension data from the Neosense measuring system, from the time points when a blood gas sample was collected, will be recorded. This data will be compared to the oxygen tension value from the blood gas sample collected at the same time point. The blood gas samples will be analysed according to clinical and laboratory routine.

The infants will remain in the study as long as the Neosense measuring system is used.

ELIGIBILITY:
Inclusion Criteria:

* Sick newborn infants where the clinical routine indicates use of an umbilical catheter. At least one of the criteria below should be fulfilled:

  * The infant needs invasive measurement of blood pressure.
  * The infant needs repetitive sampling of blood.
  * The infant needs prolonged infusion(s) > 2 days.
  * The infant needs infusion of vessel irritating and potentially vessel harming solutions.
  * The infant is born extremely preterm (before 28+0 weeks gestational age).
  * A newborn infant with severe respiratory disorder, requiring oxygen treatment (more than 40% Fraction of inspired oxygen (FiO2)).
  * The infant is undergoing therapeutic hypothermia following asphyxia ("oxygen deficiency at birth").
  * The infant has a severe infection/sepsis.
* Signed informed consent form by both parents (or guardians), (if the infant has only one parent (or guardian) one informed consent is required).

Exclusion criteria:

* Gastroschisis
* Omphalocele
* Peritonitis
* Necrotizing enterocolitis
* Omphalitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-03-06 (Actual); Study Completion 2021-03-06 (Actual)

PRIMARY OUTCOMES:
Measurement performance of an intravascular oxygen sensor in the Neosense system. | Average of measurement comparisons done at every blood gas sample, i.e. every 4th - 6th hour during the study (up to 8 days)
  The oxygen tension measured by the Neosense system, compared to the oxygen tension measured by a blood gas analyser.

SECONDARY OUTCOMES:
Clinical complications with the Neosense catheter. | During study, up to 8 days
  The number of occasions when the Neosense catheter had to be removed and the underlying reason. This includes all anticipated device effects as well as placing the catheter in the wrong vessel, impossible to measure blood pressure, collect blood samples and/or administer fluids.
Any deviations from normal procedures when inserting an umbilical catheter. | During day 1
  Number of attempts to place the catheter for each patient. Any accessories needed to introduce or handle the Neosense catheter.
Number of monitor lockups or battery depletions | During study, in average 4-5 days
  Timepoint for monitor lockup or battery depletion, in case of occurrence.
Usability and functionality of the Neosense monitor. | During study, in average 4-5 days
  Occurence of anticipated adverse device effects for the monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Mats B Blennow, MD, Prof., Principal Investigator — Karolinska University Hospital
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Huddinge
  - Uppsala University Children's Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No